CLINICAL TRIAL: NCT03818217
Title: Effects of a Socially Assistive Robot Coach on Physical and Psychosocial Outcomes of Caregivers, Dementia Trainers and Persons With Dementia Living at Home: a Mixed Method Randomized Clinical Trial
Brief Title: Effects of a Robot on Physical and Psychosocial Outcomes of Persons With Dementia and Their Social Environment at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Joanneum Research Forschungsgesellschaft mbH (Other); Sozialverein Deutschlandsberg (Unknown); Humanizing Technologies GmbH (Unknown)
Responsible Party: Principal Investigator, Sandra Schüssler, Deputy Head of the Institute of Nursing Science, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 30-401ex17/18
Record Dates: First submitted 2019-01-09; First posted 2019-01-28 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Dementia
Keywords: socially assistive robot; humanoid robot; motivation; home care; cognitive training; physical training; caregivers; dementia trainers; Computers, handheld
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Intervention group: 20 persons with dementia will receive a socially assistive humanoid robot coach (including a theratainment app for physical and cognitive exercises).
  The control group (also 20 persons with dementia) will get a Tablet training including the same theratainment app as in the intervention group, but without the robot.
Masking Description: Masking is not possible, because of the used interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coach Pepper group (Experimental): Pepper is a humanoid socially assistive robot.
  Interventions: Device: Coach Pepper group
- Tablet group (Other): Tablet training
  Interventions: Device: Tablet group

INTERVENTIONS:
Device: Coach Pepper group — Robot Pepper's height is 1.20 meters and it weighs 28 kilograms. Pepper's operation time is about 12 hours.
  Pepper will be called as Coach Pepper because s/he is virtually connected via web interfaces with a theratainment app including cognitive and physical training .
  Arms: Coach Pepper group
Device: Tablet group — The Tablet provides a theratainment app including cognitive and physical training.
  Arms: Tablet group

SUMMARY:
Background:

Dementia rates are increasing worldwide and consequently burden global healthcare resources to a serious degree. However, there is a declining number of caregivers to provide care. It is for this reason that many new technologies, such as socially assistive robots, have been developed because of their potential to support caregivers in promoting the independence of people with dementia.

Most of the (socially assistive) robots have so far been tested for people without dementia in mainly laboratory or in institutional settings, like nursing homes. Consequently, there is a lack of knowledge about the possible uses of robots from the perspective of those affected by dementia in real-life/care situations (e.g. at home). Testing in a laboratory setting cannot capture the complexity and high variability of everyday situations occurring during the care of persons with dementia.

Aim:

The aim is to investigate the effect of a socially assistive humanoid robot on the physical and psychosocial outcomes of caregivers, dementia trainers and persons with dementia living at home.

Methods:

The design is a mixed method randomized clinical trial. As an intervention, 20 persons with dementia and their relatives will receive a socially assistive humanoid robot coach (including a theratainment app for physical and cognitive exercises). The control group (also 20 persons with dementia and their relatives) will receive a tablet including the same theratainment app as in the intervention group, but without the robot.

Data will be collected using sensor data of the robot and the tablet, eye tracking, questionnaires, observation and interviews. There are also questionnaires for the relatives (n=40), dementia trainers (n=5) and professional caregivers (n=5).

Data analysis is quantitative (descriptive statistics, median regression, covariance analysis, wilcoxon rank-sum test) and qualitative (content analysis).

The planned study supports the further development of socially assistive robots with regard to the individual needs of persons with dementia living at home.

ELIGIBILITY:
Inclusion criteria:

Persons with dementia:

* adults
* living at home
* all types of dementia (except frontotemporal dementia)
* light and moderate dementia (MMSE 10 and above)
* light dementia: living alone or with relative at home (if alone: the relative should live in the neighborhood and be in daily contact with the person with dementia)
* moderate dementia: living with a relative at home
* receive professional and/or non-professional care or no care
* speak and understand German
* have no physical, auditory or visual restrictions, which would make the application of the interventions impossible.
* do not take any dementia-specific medication or have been taking dementia-specific medication for at least 3 months; condition stable and no change expected during the study period
* do not take antipsychotics and antidepressants or have been taking them for at least 14 days before study start
* children and pets in the household after previous individual discussion

Relatives:

* relatives of the participating persons with dementia (adults)
* relatives means family members, like spouse, daughter, aunt, ... or significant others like friends and neighbors
* living or not living with the person with dementia in the same household (in the case of moderate dementia, relatives must live in the same household)
* person with dementia receives or receives no professional care
* relative provides or does not provide care
* if the persons with dementia receive paid 24-hour care (regardless of whether they have mild or moderate dementia), a relative still has to be recruited as a participant (this relative must live in the same house or household and be in daily contact with the person with dementia)
* speak and understand German

Professional caregivers

* adults
* nurses or nursing assistants
* speak and understand German

Dementia trainers

* adults
* trained as M.A.S. (Morbus Alzheimer Syndrome) trainer
* train the participants with dementia at home
* speak and understand German

Exclusion criteria:

Persons with dementia:

* frontotemporal dementia
* known aggressive behavior

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change of motivation (persons with dementia) | 3 weeks
  The "Apathy Evaluation Scale" is a scale to measure motivation because apathy can be understood as a loss of motivation. The scale has 18 items (4-point Likert scale). 18-72 points can be obtained. Higher scores correspond to a higher degree of apathy and therefore lower motivation. Furthermore, sensor data of the robot Pepper/ the tablet will be analysed (usage of different functions).
Change of care burden (relatives) | 3 weeks
  The "Zarid Burden Interview" captures the subjective burden of caregivers. The instrument has 22 items (5-point Likert scale). 0 - 88 points can be obtained. Higher scores indicate greater caregiver distress.

SECONDARY OUTCOMES:
Change of quality of life (persons with dementia, relatives): The "Dementia Quality of Life Instrument" | 3 weeks
  The "Dementia Quality of Life Instrument" will be used for the participants with dementia. The instrument has 28 items (4-point Likert scale) in 5 domains (self-esteem: 4 items; positive affect/humor- 6 items, negative affect - 11 items; feelings of belonging - 3 items; sense of aesthetics - 5 items). A global quality-of-life item is also included but does not contribute to the overall score. For every item, 1 to 4 points can be obtained, with higher scores indicating better quality of life. For the relatives, the short version of the "World Health Organization Quality of Life Scale" will be used. It has 26 items and 4 domains (physical health, psychological, social relationship, environment). For every item, 1-5 points can be obtained. In general, higher domain scores indicate a higher quality of life.
Change of care dependency (persons with dementia) | 3 weeks
  The "Care Dependency Scale" has 15 items (5-point Likert scale). 15-75 points can be obtained. Lower scores indicate a higher degree of care dependency.
Change of mobility (persons with dementia) | 3 weeks
  The "Timed UP and GO Test" measures the time (in seconds) an individual needs to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down. Interpretation: <10 seconds = completely unrestricted; 10-19 seconds = less mobile, but still unrestricted; 20 - 29 seconds = limited mobility; >30 seconds = pronounced mobility restriction. 14 seconds and more has been shown to indicate a high risk of falls. Furthermore, sensor data of the robot Pepper will be analysed (activity during physical training with the theratainment app).
Change of cognition (persons with dementia) | 3 weeks
  The "Montreal Cognitive Assessment" has 30 items in 8 domains of cognitive functioning: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. 0-30 points can be obtained. Lower scores indicate a higher degree of cognitive impairment. Furthermore, sensor data of the theratainment app on the tablet will be analysed (performance of cognitive training).
Change of depression (persons with dementia, relatives) | 3 weeks
  The short version of the "Geriatric Depression Scale" will be used for persons with dementia. The scale has 15 items (yes/no answers). 0-15 points can be obtained. Higher scores indicate a higher level of depressive symptoms. The "Center for Epidemiological Studies Depression Scale" will be used for the relatives. The scale has 20 items (4-point Likert scale). 0-60 points can be obtained. Higher scores indicate a higher level of depressive symptoms.
Technology acceptance (persons with dementia, relatives, dementia trainers, professional caregivers) | 3 weeks
  The "Technology Usage Inventory" measures acceptance with 9 scales (curiosity, anxiety, interest, usability/user friendliness, immersion, utility, skepticism and accessibility, intention to use) and 30 items (7-point Likert scale). 26-182 points can be obtained (except for the scale "Intention to Use", which is a visual analogue scale with a ten-centimeter-long horizontal line with the two end-points "agree" and "disagree". A cross on the line indicates the degree of agreement. For the evaluation, the distance from the right end-point (disagreement) to the answer cross on the line is measured. This distance (in millimeters) is determined and summed up for all three items (maximum:300, Minimum:0). For all scales, higher levels on the respective scales indicate a higher level of expression in the respective construct. Additionally, individual interviews (people with dementia, relatives) and focus groups (other participants) will be conducted to obtain more in-deep knowledge
Change of usability/acceptance (persons with dementia): semi-structured observation | 3 weeks
  An open, semi-structured observation of persons with dementia interacting with the robot at home will be conducted by professional caregivers.
Change of affect (relatives) | 3 weeks
  The "Positive and Negative Affect Schedule" has 20 items (5-point Likert scale) with 2 dimensions (positive affect, negative affect). In total, 20 - 100 points can be obtained. Higher scores indicate higher positive or rather negative affect.
Change of behavioral problems (persons with dementia) | 3 weeks
  The "Neuropsychiatric Inventory (NPI)" has 12 dimensions (delusions, agitation/aggression, depression, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability, aberrant motor behavior, sleep and night-time behavior disorders, appetite and eating disorders). Each of the 12 domains is rated in terms of severity (ranging from 0 = absent to 3 = severe) and frequency (ranging from 1 = rare to 4 = frequent). The score of each item is then calculated by multiplying severity by frequency, thus obtaining a score ranging between 0 and 12. The total NPI score is finally obtained by adding all the single item scores (thus, ranging from 0 to 144). Higher scores indicate greater psychopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Schüssler, Dr., Principal Investigator — Medical Univesity of Graz, Institute of Nursing Science
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ADI. Journey of caring: an analysis of long-term care for dementia. ADI, London, 2013
- [Background] Bioethikkommission (Bioethics Commission). Roboter in der Betreuung alter Menschen - Stellungnahme der Bioethikkommission (Robots in the care of older people - statement of the Bioethics Commission). Geschäftsstelle der Bioethikkommission, Vienna, 2018
- [Background] Boman IL, Lundberg S, Starkhammar S, Nygard L. Exploring the usability of a videophone mock-up for persons with dementia and their significant others. BMC Geriatr. 2014 Apr 16;14:49. doi: 10.1186/1471-2318-14-49. PMID 24739662
- [Background] Lauriks S, Reinersmann A, Van der Roest HG, Meiland FJ, Davies RJ, Moelaert F, Mulvenna MD, Nugent CD, Droes RM. Review of ICT-based services for identified unmet needs in people with dementia. Ageing Res Rev. 2007 Oct;6(3):223-46. doi: 10.1016/j.arr.2007.07.002. Epub 2007 Aug 2. PMID 17869590
- [Background] Mao HF, Chang LH, Yao G, Chen WY, Huang WN. Indicators of perceived useful dementia care assistive technology: Caregivers' perspectives. Geriatr Gerontol Int. 2015 Aug;15(8):1049-57. doi: 10.1111/ggi.12398. Epub 2014 Nov 19. PMID 25407039
- [Background] NHI, WHO. Global Health and Aging http://www.who.int/ageing/publications/global_health.pdf. Accessed 18. Dezember 2017, 2011.
- [Background] OECD. Adressing Dementia - the OECD response. OECD publishing, Paris, 2015.
- [Background] Pino M, Boulay M, Jouen F, Rigaud AS. "Are we ready for robots that care for us?" Attitudes and opinions of older adults toward socially assistive robots. Front Aging Neurosci. 2015 Jul 23;7:141. doi: 10.3389/fnagi.2015.00141. eCollection 2015. PMID 26257646
- [Background] Prince et al. World Alzheimer Report 2016 - Improving healthcare for people living with dementia. ADI, UK, 2016
- [Background] Robert Koch Institut. Gesundheit in Deutschland. Gesundheitsberichterstattung des Bundes (Health in Germany. Health report of the federal government). Gemeinsam getragen von RKI und Destatis. RKI, Berlin, 2015
- [Background] Wang RH, Sudhama A, Begum M, Huq R, Mihailidis A. Robots to assist daily activities: views of older adults with Alzheimer's disease and their caregivers. Int Psychogeriatr. 2017 Jan;29(1):67-79. doi: 10.1017/S1041610216001435. Epub 2016 Sep 23. PMID 27660047